CLINICAL TRIAL: NCT03631979
Title: Regular Intestinal Lavage to Promote Enteral Feeding and Prevent Necrotizing Enterocolitis in Extremely Preterm Infants. A Randomized Controlled Trial Protocol
Brief Title: Intestinal Lavage to Promote Enteral Feeding and Prevent Necrotizing Enterocolitis in Extremely Preterm Infants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Spyridon Gialamas, MD, PhD, Uppsala County Council, Sweden
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018/141
Record Dates: First submitted 2018-07-13; First posted 2018-08-15 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Necrotizing Enterocolitis; Time to Full Enteral Nutrition
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Regular intestinal lavage with normal saline twice per day, starting after randomization and not later than 24 hours of age, and continued until full enteral nutrition of 170ml/kg/day is achieved or NEC diagnosis (Bell stage II or more) is established, which one comes first. The intervention will be applied at a maximum of 2 weeks from birth.
  Interventions: Other: Intestinal lavage with normal saline
- Control group (No Intervention): Current routine for extremely preterm infants that do not defecate adequately will be applied.

INTERVENTIONS:
Other: Intestinal lavage with normal saline — Specially trained pediatric surgeon will administer 10ml/kg pre-warmed (37oC) normal saline via a single-use rectal tube of size 6FR twice per day, aiming at a depth of maximum 10 cm/kg, starting after randomization and not later than 24 hours of age, and continued until full enteral nutrition of 170ml/kg/day is achieved or NEC diagnosis (Bell stage II or more) is established, which one comes first. However, the intervention will be applied at a maximum of 2 weeks from birth.
  Arms: Intervention group

SUMMARY:
Optimizing enteral nutrition (EN) is challenging in extremely preterm infants due to feeding intolerance that relates to the functional gastrointestinal immaturity. Early feeding is a safe way to promote postnatal gastrointestinal maturation and, when compared with delayed enteral feeding, provide benefit, such as reduced time to full enteral feedings (TFF) and number of parenteral nutrition (PN) days. Failure to develop oral feeding competence often leads to growth failure, longer hospital stays, dependence on PN and its complications, and influences long-term growth and developmental outcomes. Feeding with human breast milk has a protective effect against necrotizing enterocolitis (NEC) compared with formula, whereas feeding intolerance is one of the early signs of NEC. Delayed passage of meconium is a risk factor for feeding intolerance in preterm very low birth weight neonates and specific meconium microbiota characteristics have been linked to increased risk of NEC. This randomized controlled trial (RCT) aims at evaluating the effect of regular intestinal lavage using normal saline on the TFF and severe complications such as NEC and sepsis, in extremely preterm infants. Investigators aim also to follow children´s neurological development until 5,5 years of age. The study will include one intervention group of 100 subjects that will receive regular rectal washout with normal saline and equal number of control subjects, treated according to current routine. The trial is preliminarily estimated to last between year 2018 and 2022. Investigators will monitor closely for possible adverse events. The results are going to be published in reviewed medical journal.

DETAILED DESCRIPTION:
The study will be designed and conducted as a two-arm parallel, open-label, randomized controlled trial (RCT) at a tertiary-care hospital.

No masking will be applied, in order not to expose the control group to sham interventions of no benefit or potential harm.

A blinded research coordinator will randomly assign eligible infants using a computer software-based randomization system (default) or sealed, numbered, and opaque envelopes (back-up), with a 1:1 allocation ratio, as soon as possible and not later than 24 hours from birth.

Sample size calculation is based on the incidence of NEC, as the rarest of the events that will be studied, which is currently about 15% among extremely preterm infants at the investigators' unit, as mentioned above. For study power of at least 70%, confidence level of 5%, and an expected decrease of NEC incidence from 15% to 8%, each study arm should include about 100 participants. Each year, the investigators' unit treats about 70 infants born in GA 22+0 - 26+6. Supposing a participation rate of 70%, it is estimated that the recruitment period should last between 3 and 4 years, preliminarily starting during 2018. However, a recruitment period of maximum 5 years will be allowed.

Current feeding regimen and feeding intolerance guidelines will be applied for both study arms.

Intervention The following intervention will be applied to the intervention group: specially trained pediatric surgeon will administer 10ml/kg pre-warmed (37oC) normal saline via a single-use rectal tube of size 6FR twice per day, aiming at a depth of maximum 10 cm/kg, starting after randomization and not later than 24 hours of age, and continued until full enteral nutrition of 170ml/kg/day is achieved or NEC diagnosis (Bell stage II or more) is established, which one comes first. However, the intervention will be applied at a maximum of 2 weeks from birth. Besides, the intervention will be withheld in case of suspicion of infection or NEC but will be resumed if antibiotics are not introduced and discontinuation of feeds does not exceed 48 hours. Early stopping criteria include infection / sepsis or NEC suspicion necessitating prolonged discontinuation of feeds > 48 hours and / or antibiotics, circulatory instability or adverse events. The intervention will only be applied at the NICU of University Children's Hospital in Uppsala and will be discontinued if the infant is transferred to another hospital.

Standard departmental guidelines will be followed regarding ventilation, choice of PN, invasive monitoring, and management of sepsis and/or necrotizing enterocolitis (NEC) for both the intervention and the control groups.

Comparison group

The following guidelines are currently applied at the investigators' unit for extremely preterm infants that do not defecate adequately:

If the child has not passed meconium or has already passed meconium / feces but has not defecated for 3-4 days:

* If there are no symptoms: continued EN, follow-up of clinical status and defecation pattern. If the child has not defecated for another 1-2 days (and remains asymptomatic), consider the following treatment strategy to facilitate defecation:

  1. Tactile perineal stimulation is performed by a nurse, using a room temperature damp compress
  2. Cautious rectal stimulation is performed by a nurse, using a rectal catheter size 6FR; depth 1 - 2 cm
  3. Step 1 & 2 is repeated depending on effect and defecation pattern
  4. If Step 1 & 2 does not result in defecation and the clinical status is unchanged, enema with 4mL / kg sodium chloride 9mg / mL is given
  5. In case of no effect, a pediatric surgeon is consulted, and consideration is given to continued treatment; (1) watchful waiting alternatively repeated enema (2) rectal washout with 10 mL / kg sodium chloride 9mg / mL (3) further radiological and laboratory investigations
* In case of symptoms (cardiorespiratory instability, impaired abdominal status, vomiting, bilious residuals, etc.): EN is withheld, pediatric surgeon is consulted and radiological / laboratory investigations as well as early treatment with antibiotics (tazobactam / piperacillin + gentamicin) is considered.

Follow-up All extremely preterm infants hospitalized in the investigators' unit are discharged home at about GA 35+0. Infants regionally belonging to another hospital are usually transferred to the "home hospital unit" not earlier than GA 28+0. After hospital discharge, all extremely preterm infants are routinely followed-up according to a nationwide schedule, until the age of 5,5 years. Data mostly concerning children's growth as well as neurological and psychomotor development are collected, and interventions are made as needed.

Study participants will be followed-up until full term corrected age (GA 40 +0), and medical information including possible treatments as well as diagnosis of NEC or other gastrointestinal complication, sepsis, PDA, BPD, ROP, IVH, hyperbilirubinemia, growth parameters (weight, length, head circumference) and mortality will be collected by the investigators from the treating physicians and electronic medical records. All the clinical, laboratory and radiological findings of infants treated at the investigators' unit are routinely and continuously registered in detail, with the use of medical computer software, during the whole hospitalization period, and these data will be readily accessible to the investigators. Besides, data on children's growth and neurological development will be collected from the electronic medical records, until the age of 5,5 years. The above-mentioned data of study participants that have been transferred to the home or other hospital unit will be collected by the investigators though communication with the treating physician at the respective hospital.

Documentation All data relevant to the study collected by the investigators will be registered and de-identified in electronic database with password-protected access allowed only to the investigators.

Refuse to enrollment and subject dropouts Refusals to enroll the study and dropouts of the study and the respective reasons will be documented and reported in the results. Effort will be made to replace each of these subjects with another infant of the same gestational age.

Completion of the study The study will be completed when the number of 100 subjects per study arm is reached (a maximum of 130 subjects per study arm will be allowed), estimated to be achieved by the year 2022 (and not later than year 2023).

Statistical analysis Numerical data with a gaussian distribution will be expressed as means (standard deviation), otherwise as medians (ranges). Anderson-Darling test will be used to assess the normality of the data. Numerical values will be compared between intervention and control groups using t-tests or the Mann-Whitney U test. Categorical variables will be compared using χ2 or Fisher's exact tests. Times to achieve full enteral feeding will be compared by the log rank test. Multiple Cox regression analysis will be used to adjust for covariates, such as gestational age and birth weight. IBM SPPS software (current version at the time of publication) will be used for all calculations and a p-value of <0,05 will be considered significant.

Interim analysis will be conducted when 35 infants have been recruited in each study arm (estimated about 1,5 years from study start). Another interim analysis will be conducted when 65 infants have been recruited in each study arm (estimated about 3 years from study start). Unplanned interim analysis will also be conducted in case of subjectively estimated too obvious difference between the groups regarding the primary outcomes, at any time during the study. The study will be discontinued as soon as an interim analysis shows statistically significant results regarding the primary outcomes or severe adverse events.

Ethical considerations The study protocol will be submitted for approval to the Regional Ethical Review Board in Uppsala and subsequently registered at the international registry of clinical trials, ClinicalTrials.gov. The parents of the infants will be informed about the study by specially trained personnel, both verbally and in writing, before the child is born or, whenever that is not possible, as soon as possible after birth. Upon agreement to participate, written informed consent will be obtained from the parents, before enrollment in the study. Additionally, the parents will be clearly informed about the possibility to leave the study any time they wish.

None of the studies published so far reported any adverse events by induced meconium evacuation, with the exception of a higher proportion of NEC (although not statistically significant), vomiting, nausea and bradycardia with the use of oral gastrografin, and a non-significant trend towards increased risk of NEC with the use of glycerine enemas or suppositories compared with no treatment. However, in the RCT study described herein, both health personnel involved in the participating infants' daily care and the investigators are going to closely monitor for possible adverse events. Possible adverse events could be: rectal bleeding (including occult rectal bleeding-induced anemia), fluid loss due to overstimulation of immature intestines of preterm infants or the opposite effect, namely intestinal absorption of given saline, leading to hypervolemia and electrolyte disturbances, mainly hyponatremia. A safety monitoring committee will monitor adverse events with predefined stopping rules. Early stopping criteria will be applied in case of medical instability, as mentioned above. Furthermore, the whole study will be discontinued in case of too obvious positive effect, making it unethical to deprive the control group of the intervention, or in case of severe adverse events.

The inclusion of study participants in other interventional studies could intervene with the outcomes intended to be investigated in the study herein, rendering it difficult to retrieve definitive conclusions. Thus, study participants will not be included in other interventional studies at the same time.

The intervention will be discontinued if the infant is transferred to another hospital, as mentioned before. The decision to transfer a study subject to home or other hospital unit will only be based on current criteria and will not be affected by the participation in the study. Study participation is not expected to delay the transfer to home hospital and prolong the stay at our NICU in Uppsala, unless a severe adverse event should occur.

Reporting and dissemination Following the study, data will be analysed by the research group and the results will be published in reviewed medical journals and possibly presented in a neonatology conference, hopefully during year 2023. It is difficult to provide a precise time schedule. Patient data collection is estimated to last about 4 years. Data analysis thereafter is time consuming and may last one more year until the whole project is completed and ready for publication. All the principal investigators will have free access to raw data and the right to publication.

ELIGIBILITY:
Inclusion Criteria:

* born at Akademiska hospital in Uppsala
* gestational age between 22 weeks + 0 days and 26 weeks +6 days
* written informed consent obtained from both guardians before enrollment in the study.

Exclusion Criteria:

* major dysmorphic features consistent with chromosomal abnormality
* major congenital anomalies, such as gastrointestinal disorders
* circulatory instability during the first hours of life

Ages: 22 Weeks to 26 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2031-11 (Estimated)

PRIMARY OUTCOMES:
Time to full enteral nutrition (FEN) | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  The time period between birth and achievement of enteral nutrition of 170ml/kg/d (days)

SECONDARY OUTCOMES:
Necrotizing enterocolitis (NEC) | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  Incidence of NEC
Neonatal sepsis | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  Incidence of neonatal sepsis
Incidence of Retinopathy of Prematurity (ROP) | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  Incidence of ROP
Grade of ROP | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  According to the International Classification of ROP (Arch Ophthalmol. 2005)
Bronchopulmonary dysplasia (BPD) | From birth until 36 weeks postnatal age or discharge, whichever comes first
  Incidence of BPD
Severity of BPD | From birth until 36 weeks postnatal age or discharge, whichever comes first
  According to NICHD/NHLBI/ORD guidelines (Am J Respir Crit Care Med. 2001)
Incidence of Intraventricular Hemorrhage (IVH) | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  Incidence of IVH
Grade of IVH | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  According to Papile's classification
Incidence of Patent Ductus Arteriosus (PDA) | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  Incidence of PDA
Hemodynamic significance of PDA | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  Based on echocardiographic assessment
Time to regain birth weight (BW) | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  The time period between birth and regaining of BW (days)
Growth (weight) | From birth until the age of 5,5 years
  Z-score of weight in kilograms
Growth (length) | From birth until the age of 5,5 years
  Z-score of length in cm
Growth (head circumference) | From birth until the age of 5,5 years
  Z-score of head circumference in cm
Mortality | From birth until 5,5 years of age
  Mortality
Duration of hospital stay | From birth until the age of 1 year
  Age of the child at the time of hospital discharge (days)
Duration of parenteral nutrition (PN) | From birth until full term corrected age (gestational age 40 weeks + 0 days) or hospital discharge, whichever comes first
  Number of days on PN (days)
Neurological development | From birth until 5,5 years age
  Assessed according to the national program for follow up of extremely preterm infants in Sweden. Assessments include examination by neonatologist, pediatric neurologist, psychologist, physiotherapist, audiologist, opthalmologist, at prespecified intervals until the age of 5,5 years
Intestinal failure-associated liver disease (IFALD) | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  Incidence of IFALD
Incidence of hyperbilirubinemia | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  Incidence of hyperbilirubinemia
Severity of hyperbilirubinemia | From birth until full term corrected age (gestational age 40 weeks + 0 days)
  Maximum serum level of unconjugated and conjugated bilirubin (μmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Normann, Chair, Study Chair — Neonatal Intensive Care Unit, Akademiska Hospital; Spyridon Gialamas, MD, PhD, Principal Investigator — Neonatal Intensive Care Unit, Akademiska Hospital
Locations (1):
- Neonatal intensiv care unit, 95F, Akademiska hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deshmukh M, Balasubramanian H, Patole S. Meconium Evacuation for Facilitating Feed Tolerance in Preterm Neonates: A Systematic Review and Meta-Analysis. Neonatology. 2016;110(1):55-65. doi: 10.1159/000444075. Epub 2016 Apr 7. PMID 27050644
- [Background] Park J, Knafl G, Thoyre S, Brandon D. Factors associated with feeding progression in extremely preterm infants. Nurs Res. 2015 May-Jun;64(3):159-67. doi: 10.1097/NNR.0000000000000093. PMID 25932696
- [Background] Morgan J, Young L, McGuire W. Delayed introduction of progressive enteral feeds to prevent necrotising enterocolitis in very low birth weight infants. Cochrane Database Syst Rev. 2014;2014(12):CD001970. doi: 10.1002/14651858.CD001970.pub5. Epub 2014 Dec 1. PMID 25436902
- [Background] Culpepper C, Hendrickson K, Marshall S, Benes J, Grover TR. Implementation of Feeding Guidelines Hastens the Time to Initiation of Enteral Feeds and Improves Growth Velocity in Very Low Birth-Weight Infants. Adv Neonatal Care. 2017 Apr;17(2):139-145. doi: 10.1097/ANC.0000000000000347. PMID 27750266
- [Background] Klein CJ, Revenis M, Kusenda C, Scavo L. Parenteral nutrition-associated conjugated hyperbilirubinemia in hospitalized infants. J Am Diet Assoc. 2010 Nov;110(11):1684-95. doi: 10.1016/j.jada.2010.08.012. PMID 21034882
- [Background] Nehra D, Fallon EM, Puder M. The prevention and treatment of intestinal failure-associated liver disease in neonates and children. Surg Clin North Am. 2011 Jun;91(3):543-63. doi: 10.1016/j.suc.2011.02.003. Epub 2011 Apr 15. PMID 21621695
- [Background] Embleton ND, Simmer K. Practice of parenteral nutrition in VLBW and ELBW infants. World Rev Nutr Diet. 2014;110:177-89. doi: 10.1159/000358466. Epub 2014 Apr 11. PMID 24751629
- [Background] Lauriti G, Zani A, Aufieri R, Cananzi M, Chiesa PL, Eaton S, Pierro A. Incidence, prevention, and treatment of parenteral nutrition-associated cholestasis and intestinal failure-associated liver disease in infants and children: a systematic review. JPEN J Parenter Enteral Nutr. 2014 Jan;38(1):70-85. doi: 10.1177/0148607113496280. Epub 2013 Jul 26. PMID 23894170
- [Background] Maisels MJ. Managing the jaundiced newborn: a persistent challenge. CMAJ. 2015 Mar 17;187(5):335-43. doi: 10.1503/cmaj.122117. Epub 2014 Nov 10. No abstract available. PMID 25384650
- [Background] Patel AL, Kim JH. Human milk and necrotizing enterocolitis. Semin Pediatr Surg. 2018 Feb;27(1):34-38. doi: 10.1053/j.sempedsurg.2017.11.007. Epub 2017 Nov 6. PMID 29275815
- [Background] Gephart SM, McGrath JM, Effken JA, Halpern MD. Necrotizing enterocolitis risk: state of the science. Adv Neonatal Care. 2012 Apr;12(2):77-87; quiz 88-9. doi: 10.1097/ANC.0b013e31824cee94. PMID 22469959
- [Background] Leach ST, Lui K, Naing Z, Dowd SE, Mitchell HM, Day AS. Multiple Opportunistic Pathogens, but Not Pre-existing Inflammation, May Be Associated with Necrotizing Enterocolitis. Dig Dis Sci. 2015 Dec;60(12):3728-34. doi: 10.1007/s10620-015-3830-6. Epub 2015 Aug 7. PMID 26250832
- [Background] Kessmann J. Hirschsprung's disease: diagnosis and management. Am Fam Physician. 2006 Oct 15;74(8):1319-22. PMID 17087425
- [Background] Meetze WH, Palazzolo VL, Bowling D, Behnke M, Burchfield DJ, Neu J. Meconium passage in very-low-birth-weight infants. JPEN J Parenter Enteral Nutr. 1993 Nov-Dec;17(6):537-40. doi: 10.1177/0148607193017006537. PMID 8301808
- [Background] Verma A, Dhanireddy R. Time of first stool in extremely low birth weight (< or = 1000 grams) infants. J Pediatr. 1993 Apr;122(4):626-9. doi: 10.1016/s0022-3476(05)83550-4. PMID 8463914
- [Background] Ibrahim T, Li Wei C, Bautista D, Sriram B, Xiangzhen Fay L, Rajadurai VS. Saline Enemas versus Glycerin Suppositories to Promote Enteral Feeding in Premature Infants: A Pilot Randomized Controlled Trial. Neonatology. 2017;112(4):347-353. doi: 10.1159/000477999. Epub 2017 Aug 3. PMID 28768263
- [Background] Shim SY, Kim HS, Kim DH, Kim EK, Son DW, Kim BI, Choi JH. Induction of early meconium evacuation promotes feeding tolerance in very low birth weight infants. Neonatology. 2007;92(1):67-72. doi: 10.1159/000100804. Epub 2007 Mar 14. PMID 17356305
- [Background] Shinde S, Kabra NS, Sharma SR, Avasthi BS, Ahmed J. Glycerin suppository for promoting feeding tolerance in preterm very low birthweight neonates: a randomized controlled trial. Indian Pediatr. 2014 May;51(5):367-70. doi: 10.1007/s13312-014-0418-8. PMID 24953576
- [Background] Khadr SN, Ibhanesebhor SE, Rennix C, Fisher HE, Manjunatha CM, Young D, Abara RC. Randomized controlled trial: impact of glycerin suppositories on time to full feeds in preterm infants. Neonatology. 2011;100(2):169-76. doi: 10.1159/000323964. Epub 2011 Apr 1. PMID 21455007
- [Background] Haiden N, Jilma B, Gerhold B, Klebermass K, Prusa AR, Kuhle S, Rohrmeister K, Kohlhauser-Vollmuth C, Pollak A. Small volume enemas do not accelerate meconium evacuation in very low birth weight infants. J Pediatr Gastroenterol Nutr. 2007 Feb;44(2):270-3. doi: 10.1097/MPG.0b013e31802c685a. PMID 17255844
- [Background] Mena N P, Leon Del P J, Sandino P D, Ralmolfo B P, Sabatelli D, Llanos M A, Milet L B. [Meconium evacuation to improve feeding tolerance in very low birth weight preterm infants (Emita Protocol)]. Rev Chil Pediatr. 2014 Jun;85(3):304-11. doi: 10.4067/S0370-41062014000300006. Spanish. PMID 25697247
- [Background] Saenz de Pipaon Marcos M, Teresa Montes Bueno M, Sanjose B, Gil M, Parada I, Amo P. Randomized controlled trial of prophylactic rectal stimulation and enemas on stooling patterns in extremely low birth weight infants. J Perinatol. 2013 Nov;33(11):858-60. doi: 10.1038/jp.2013.86. Epub 2013 Aug 1. PMID 23907087
- [Background] Anabrees J, Shah VS, AlOsaimi A, AlFaleh K. Glycerin laxatives for prevention or treatment of feeding intolerance in very low birth weight infants. Cochrane Database Syst Rev. 2015 Sep 30;2015(9):CD010464. doi: 10.1002/14651858.CD010464.pub2. PMID 26421424
- [Background] Livingston MH, Shawyer AC, Rosenbaum PL, Williams C, Jones SA, Walton JM. Glycerin enemas and suppositories in premature infants: a meta-analysis. Pediatrics. 2015 Jun;135(6):1093-106. doi: 10.1542/peds.2015-0143. Epub 2015 May 18. PMID 25986027
- [Background] Kamphorst K, Sietsma Y, Brouwer AJ, Rood PJ, van den Hoogen A. Enemas, suppositories and rectal stimulation are not effective in accelerating enteral feeding or meconium evacuation in low-birthweight infants: a systematic review. Acta Paediatr. 2016 Nov;105(11):1280-1287. doi: 10.1111/apa.13540. Epub 2016 Sep 8. PMID 27506482
- [Background] Srinivasjois R, Sharma A, Shah P, Kava M. Effect of induction of meconium evacuation using per rectal laxatives on neonatal hyperbilirubinemia in term infants: a systematic review of randomized controlled trials. Indian J Med Sci. 2011 Jul;65(7):278-85. PMID 23422701

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT03631979/Prot_SAP_000.pdf
  • Informed Consent Form (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/79/NCT03631979/ICF_001.pdf